CLINICAL TRIAL: NCT06433271
Title: Comparative Effectiveness of Transdiagnostic Behavior Therapy Vs TAU for Adjustment Disorder Following Traumatic Event Exposure
Brief Title: Transdiagnostic Behavior Therapy Vs TAU for Adjustment Disorder Following Traumatic Event Exposure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Ralph H. Johnson VA Medical Center (U.S. Federal Agency); U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ronald E. Acierno, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00134707; PR230007 (Other Grant/Funding Number: United States Army Medical Research and Development Command)
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Adjustment Disorders; Mental Disorder
Keywords: Veterans; Military Personnel
MeSH Terms: conditions — Adjustment Disorders; Mental Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transdiagnostic Behavior Therapy (TBT) (Experimental): Participants will receive 6, 30-45-minute, manualized, individual therapy sessions.
  Interventions: Behavioral: Transdiagnostic Behavior Therapy (TBT)
- Active Comparator: Treatment as Usual-Problem Solving Therapy (TAU-PST) (Active Comparator): Participants will receive 6, 30-45-minute, manualized, individual therapy sessions.
  Interventions: Behavioral: Treatment as Usual-Problem Solving Therapy (TAU-PST)

INTERVENTIONS:
Behavioral: Transdiagnostic Behavior Therapy (TBT) — TBT manualized treatment incorporates daily exposure exercises from up to four categories of avoidance that are most characteristic of the emotional disorders (i.e., situational, interoceptive, imaginal, and positive emotional).
  Arms: Transdiagnostic Behavior Therapy (TBT)
Behavioral: Treatment as Usual-Problem Solving Therapy (TAU-PST) — PST is an evidence- based psychotherapy implemented in VA Primary Care - Mental Health Integration (PC-MHI), with hundreds of VA providers trained in the intervention nationally. The primary aim of PST is to improve a patient's ability to cope with stressful events by adopting an adaptive perspective to stressors and using goal-focused, problem-solving behaviors to manage the problems associated with the stressors.
  Other Names: Moving Forward Problem Solving Therapy
  Arms: Active Comparator: Treatment as Usual-Problem Solving Therapy (TAU-PST)

SUMMARY:
Adjustment Disorder (AjD) is the most common mental health condition diagnosed in Active Duty personnel, and is diagnosed following an extreme stress event such as traumatic loss of a comrade, serious accident or injury, or other intense stress event. Despite its high prevalence, no evidence based treatment for AjD has been subjected to randomized controlled trials. This study seeks to build on the research team's pilot work across several disorders study to benefit service members and Veterans with AjD, a highly prevalent but frequently inadequately treated condition.

The investigators will compare the effects of Transdiagnostic Behavior Therapy (TBT) vs treatment as usual which is Moving Forward Problem Solving Therapy (TAU-PST) on AjD symptom outcomes. The investigators hypothesize that TBT will result in greater overall symptom reduction compared to TAU-PST.

DETAILED DESCRIPTION:
Adjustment Disorder (AjD) is the most common mental health condition diagnosed in Active Duty personnel, and is diagnosed following an extreme stress event such as traumatic loss of a comrade, serious accident or injury, or other intense stress event. Despite its high prevalence, no evidence based treatment for AjD has been subjected to randomized controlled trials.

Currently, the VA suggests a problem solving cognitive behavioral therapy, but this recommendation is not based on replicated, randomized controlled trials. Transdiagnostic Behavior Therapy (TBT), is based on key 'active components' of existing evidence based treatments such as Prolonged Exposure and Behavioral Activation, has been designed by this research team to be easily trained and inexpensively disseminated, and has been evaluated in a series of pilots with anxiety and depression disorders that, importantly, represent the key symptom classes of adjustment disorder.

Thus, the rationale for the proposed trial is that the research team has done preliminary efficacy testing of an easily exportable intervention that has impact on the key symptoms of adjustment disorder, and the standard of evidence demands replicated, randomized controlled trials to determine if initial signals of positive effect are sustained.

The study will use a 2 group repeated measures randomized controlled design to evaluate effectiveness of TBT for AjD compared to treatment as usual (TAU-PST). Participants will be randomly assigned in equal numbers (n = 75; N = 150) to one of two treatment arms: (1) TBT or (2) TAU-PST. Participants assigned to TBT will receive 6, 30-45-minute, manualized, individual therapy sessions. Participants assigned to TAU-PST will receive 6, 30-45-minute sessions of Problem-Solving Therapy. Dependent measures will include Department of Defense (DoD) specified common data elements and specific measures of AjD, PTSD, anxiety, depression, and functioning collected by blinded assessors at baseline, post-treatment, 3-month, and 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female over the age of 18 that has served, or is currently serving, in the military.
* Stable psychotropic medication for at least 4 weeks if applicable
* Current DSM-5 diagnosis of Adjustment Disorder

Exclusion Criteria:

* Active psychosis
* Suicidal ideation with clear intent
* Severe substance use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Adjustment Disorder New Module Self Report | Baseline
  The Adjustment Disorder New Module (ADNM) is a 20-item self-report measure of AjD that first asks participants to select from a list of past year stressors and to identify which was the most prominent or distressing. The second section comprises 20 items, which form six subscales in accordance with International Classification of Diseases 11th Revision (ICD-11) criteria relating to pre-occupation, failure to adapt, avoidance, depressive mood, anxiety, and impulse disturbance (Lorenz et al., 2016). Participants rate on a 4-point Likert scale how often they have experienced particular symptoms during the past two weeks, and overall symptom severity is calculated as a sum of all item scores. Total score ranges from 20-80, with a higher score indicating a higher risk of developing adjustment disorder.
Adjustment Disorder New Module Self Report | 1 week post treatment
  The ADNM is a 20-item self-report measure of AjD that first asks participants to select from a list of past year stressors and to identify which was the most prominent or distressing. The second section comprises 20 items, which form six subscales in accordance with ICD-11 criteria relating to pre-occupation, failure to adapt, avoidance, depressive mood, anxiety, and impulse disturbance (Lorenz et al., 2016). Participants rate on a 4-point Likert scale how often they have experienced particular symptoms during the past two weeks, and overall symptom severity is calculated as a sum of all item scores. Total score ranges from 20-80, with a higher score indicating a higher risk of developing adjustment disorder.
Adjustment Disorder New Module Self Report | 3 months post treatment
  The ADNM is a 20-item self-report measure of AjD that first asks participants to select from a list of past year stressors and to identify which was the most prominent or distressing. The second section comprises 20 items, which form six subscales in accordance with ICD-11 criteria relating to pre-occupation, failure to adapt, avoidance, depressive mood, anxiety, and impulse disturbance (Lorenz et al., 2016). Participants rate on a 4-point Likert scale how often they have experienced particular symptoms during the past two weeks, and overall symptom severity is calculated as a sum of all item scores. Total score ranges from 20-80, with a higher score indicating a higher risk of developing adjustment disorder.
Adjustment Disorder New Module Self Report | 6 months post treatment
  The ADNM is a 20-item self-report measure of AjD that first asks participants to select from a list of past year stressors and to identify which was the most prominent or distressing. The second section comprises 20 items, which form six subscales in accordance with ICD-11 criteria relating to pre-occupation, failure to adapt, avoidance, depressive mood, anxiety, and impulse disturbance (Lorenz et al., 2016). Participants rate on a 4-point Likert scale how often they have experienced particular symptoms during the past two weeks, and overall symptom severity is calculated as a sum of all item scores. Total score ranges from 20-80, with a higher score indicating a higher risk of developing adjustment disorder.
Generalized Anxiety Disorder Questionnaire - 7 | Baseline
  The Generalized Anxiety Disorder Questionnaire (GAD-7; Spitzer et al., 2006) consists of seven items measuring worry and anxiety symptoms. Each item is scored on a four-point Likert scale (0-3) with total scores ranging from 0 to 21 with higher scores reflecting greater anxiety severity.of Mental Disorders, Fifth Edition (DSM-5) (PCL-5) (Weathers et al., 2013) is structured to correspond to the DSM-5 PTSD criteria. The 20-items are scored on a 0-4 Likert scale for each symptom corresponding to "Not at all" to "Extremely". Total score ranges from 0 to 80, with a higher score indicating greater PTSD symptom severity.
Generalized Anxiety Disorder Questionnaire - 7 | 1 week post treatment
  The Generalized Anxiety Disorder Questionnaire (GAD-7; Spitzer et al., 2006) consists of seven items measuring worry and anxiety symptoms. Each item is scored on a four-point Likert scale (0-3) with total scores ranging from 0 to 21 with higher scores reflecting greater anxiety severity.of Mental Disorders, Fifth Edition (DSM-5) (PCL-5) (Weathers et al., 2013) is structured to correspond to the DSM-5 PTSD criteria. The 20-items are scored on a 0-4 Likert scale for each symptom corresponding to "Not at all" to "Extremely". Total score ranges from 0 to 80, with a higher score indicating greater PTSD symptom severity.
Generalized Anxiety Disorder Questionnaire - 7 | 3 months post treatment
  The Generalized Anxiety Disorder Questionnaire (GAD-7; Spitzer et al., 2006) consists of seven items measuring worry and anxiety symptoms. Each item is scored on a four-point Likert scale (0-3) with total scores ranging from 0 to 21 with higher scores reflecting greater anxiety severity.of Mental Disorders, Fifth Edition (DSM-5) (PCL-5) (Weathers et al., 2013) is structured to correspond to the DSM-5 PTSD criteria. The 20-items are scored on a 0-4 Likert scale for each symptom corresponding to "Not at all" to "Extremely". Total score ranges from 0 to 80, with a higher score indicating greater PTSD symptom severity.
Generalized Anxiety Disorder Questionnaire - 7 | 6 months post treatment
  The Generalized Anxiety Disorder Questionnaire (GAD-7; Spitzer et al., 2006) consists of seven items measuring worry and anxiety symptoms. Each item is scored on a four-point Likert scale (0-3) with total scores ranging from 0 to 21 with higher scores reflecting greater anxiety severity.of Mental Disorders, Fifth Edition (DSM-5) (PCL-5) (Weathers et al., 2013) is structured to correspond to the DSM-5 PTSD criteria. The 20-items are scored on a 0-4 Likert scale for each symptom corresponding to "Not at all" to "Extremely". Total score ranges from 0 to 80, with a higher score indicating greater PTSD symptom severity.
Patient Health Questionnaire-9 | Baseline
  The Patient Health Questionnaire-9 (PHQ-9) (Kroenke et al., 2001) is a widely used, well-validated measure of depression severity with high internal consistency (alpha .83 to .92; Cameron et al, 2008) and is correlated strongly with other depression measures. Its nine items assess affective and somatic symptoms and correspond to diagnostic criteria for major depressive disorder (MDD). This measure will also be collected every other week during treatment. Total score ranges from 0 to 27 (scores of 5-9 are classified as mild depression; 10-14 as moderate depression; 15-19 as moderately severe depression; ≥ 20 as severe depression).
Patient Health Questionnaire-9 | 1 week post treatment
  The PHQ-9 (Kroenke et al., 2001) is a widely used, well-validated measure of depression severity with high internal consistency (alpha .83 to .92; Cameron et al, 2008) and is correlated strongly with other depression measures. Its nine items assess affective and somatic symptoms and correspond to diagnostic criteria for MDD. This measure will also be collected every other week during treatment. Total score ranges from 0 to 27 (scores of 5-9 are classified as mild depression; 10-14 as moderate depression; 15-19 as moderately severe depression; ≥ 20 as severe depression).
Patient Health Questionnaire-9 | 3 months post treatment
  The PHQ-9 (Kroenke et al., 2001) is a widely used, well-validated measure of depression severity with high internal consistency (alpha .83 to .92; Cameron et al, 2008) and is correlated strongly with other depression measures. Its nine items assess affective and somatic symptoms and correspond to diagnostic criteria for MDD. This measure will also be collected every other week during treatment. Total score ranges from 0 to 27 (scores of 5-9 are classified as mild depression; 10-14 as moderate depression; 15-19 as moderately severe depression; ≥ 20 as severe depression).
Patient Health Questionnaire-9 | 6 months post treatment
  The PHQ-9 (Kroenke et al., 2001) is a widely used, well-validated measure of depression severity with high internal consistency (alpha .83 to .92; Cameron et al, 2008) and is correlated strongly with other depression measures. Its nine items assess affective and somatic symptoms and correspond to diagnostic criteria for MDD. This measure will also be collected every other week during treatment. Total score ranges from 0 to 27 (scores of 5-9 are classified as mild depression; 10-14 as moderate depression; 15-19 as moderately severe depression; ≥ 20 as severe depression).

SECONDARY OUTCOMES:
Insomnia Severity Index | Baseline
  The Insomnia Severity Index (ISI) self-report measure captures a respondent's perception of his or her current insomnia. The ISI includes seven items that assess severity of sleep onset, sleep maintenance, and early morning awakening problems; sleep dissatisfaction; interference of sleep difficulties with daytime functioning; noticeability of sleep problems by others; and distress caused by the sleep difficulties. Each item is rated on a 4-point Likert scale and the total score ranges from 0 to 28. A higher score suggests more severe insomnia.
Insomnia Severity Index | 1 week post treatment
  The ISI self-report measure captures a respondent's perception of his or her current insomnia. The ISI includes seven items that assess severity of sleep onset, sleep maintenance, and early morning awakening problems; sleep dissatisfaction; interference of sleep difficulties with daytime functioning; noticeability of sleep problems by others; and distress caused by the sleep difficulties. Each item is rated on a 4-point Likert scale and the total score ranges from 0 to 28. A higher score suggests more severe insomnia.
Insomnia Severity Index | 3 months post treatment
  The ISI self-report measure captures a respondent's perception of his or her current insomnia. The ISI includes seven items that assess severity of sleep onset, sleep maintenance, and early morning awakening problems; sleep dissatisfaction; interference of sleep difficulties with daytime functioning; noticeability of sleep problems by others; and distress caused by the sleep difficulties. Each item is rated on a 4-point Likert scale and the total score ranges from 0 to 28. A higher score suggests more severe insomnia.
Insomnia Severity Index | 6 months post treatment
  The ISI self-report measure captures a respondent's perception of his or her current insomnia. The ISI includes seven items that assess severity of sleep onset, sleep maintenance, and early morning awakening problems; sleep dissatisfaction; interference of sleep difficulties with daytime functioning; noticeability of sleep problems by others; and distress caused by the sleep difficulties. Each item is rated on a 4-point Likert scale and the total score ranges from 0 to 28. A higher score suggests more severe insomnia.
Medical Outcome Study Short Form-36 Health Survey | Baseline
  The Short Form-36 (SF-36) (Ware & Sherbourne, 1992) is a 36-item questionnaire that measures health status, social support, and functioning over the past four weeks. Total score ranges from 0 to 100, with a higher score indicating better health status.
Medical Outcome Study Short Form-36 Health Survey | 1 week post treatment
  The SF-36 (Ware & Sherbourne, 1992) is a 36-item questionnaire that measures health status, social support, and functioning over the past four weeks. Total score ranges from 0 to 100, with a higher score indicating better health status.
Medical Outcome Study Short Form-36 Health Survey | 3 months post treatment
  The SF-36 (Ware & Sherbourne, 1992) is a 36-item questionnaire that measures health status, social support, and functioning over the past four weeks. Total score ranges from 0 to 100, with a higher score indicating better health status.
Medical Outcome Study Short Form-36 Health Survey | 6 months post treatment
  The SF-36 (Ware & Sherbourne, 1992) is a 36-item questionnaire that measures health status, social support, and functioning over the past four weeks. Total score ranges from 0 to 100, with a higher score indicating better health status.
Dose Received | 14 weeks after treatment starts
  Number of treatment sessions completed.

CONTACTS AND LOCATIONS:
Overall Officials: Ron Acierno, PhD, Principal Investigator — McGovern Medical School at UTHealth Houston
Locations (1):
- Ralph H. Johnson VA Health Care System, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gros DF. Development and initial evaluation of Transdiagnostic Behavior Therapy (TBT) for veterans with affective disorders. Psychiatry Res. 2014 Dec 15;220(1-2):275-82. doi: 10.1016/j.psychres.2014.08.018. Epub 2014 Aug 15. PMID 25193379
- [Background] Gros DF, Allan NP. A randomized controlled trial comparing Transdiagnostic Behavior Therapy (TBT) and behavioral activation in veterans with affective disorders. Psychiatry Res. 2019 Nov;281:112541. doi: 10.1016/j.psychres.2019.112541. Epub 2019 Aug 29. PMID 31514043
- [Background] Gros DF, Merrifield C, Rowa K, Szafranski DD, Young L, McCabe RE. A Naturalistic Comparison of Group Transdiagnostic Behaviour Therapy (TBT) and Disorder-Specific Cognitive Behavioural Therapy Groups for the Affective Disorders. Behav Cogn Psychother. 2019 Jan;47(1):39-51. doi: 10.1017/S1352465818000309. Epub 2018 May 29. PMID 29807553
- [Background] Gros DF, Szafranski DD, Shead SD. A real world dissemination and implementation of Transdiagnostic Behavior Therapy (TBT) for veterans with affective disorders. J Anxiety Disord. 2017 Mar;46:72-77. doi: 10.1016/j.janxdis.2016.04.010. Epub 2016 Apr 27. PMID 27158076